CLINICAL TRIAL: NCT00253552
Title: A Pilot Study of Using Filgrastim-Primed Bone Marrow in Human Leukocyte Antigen (HLA) Matched Related Donor Allogenetic Bone Marrow Transplantation for Patients With Hematologic Malignancies and Non-Malignancies
Brief Title: G-CSF-Treated Donor Bone Marrow Transplant in Treating Patients With Hematologic Disorders
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated at request of PI as study was outdated.
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000445188; OHSU-HEM-04007-L (Other: OHSU Knight Cancer Institute); OHSU-1381 (Other: OHSU IRB)
Record Dates: First submitted 2005-11-11; First posted 2005-11-15 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2010-06

CONDITIONS: Chronic Myeloproliferative Disorders; Graft Versus Host Disease; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases; Sarcoma
Keywords: graft versus host disease; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); accelerated phase chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; atypical chronic myeloid leukemia; blastic phase chronic myelogenous leukemia; childhood acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood chronic myelogenous leukemia; chronic eosinophilic leukemia; chronic idiopathic myelofibrosis; chronic myelomonocytic leukemia; chronic neutrophilic leukemia; chronic phase chronic myelogenous leukemia; de novo myelodysplastic syndromes; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; juvenile myelomonocytic leukemia; myelodysplastic/myeloproliferative disease, unclassifiable; nodal marginal zone B-cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; previously treated myelodysplastic syndromes; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; recurrent adult Burkitt lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent/refractory childhood Hodgkin lymphoma; recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood rhabdomyosarcoma; recurrent childhood small noncleaved cell lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent small lymphocytic lymphoma; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; refractory multiple myeloma; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; secondary myelodysplastic syndromes; splenic marginal zone lymphoma; stage I multiple myeloma; stage II multiple myeloma; stage III adult Burkitt lymphoma; stage III adult Hodgkin lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III chronic lymphocytic leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III multiple myeloma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV chronic lymphocytic leukemia; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; childhood myelodysplastic syndromes
MeSH Terms: conditions — Myeloproliferative Disorders; Graft vs Host Disease; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Sarcoma; Congenital Abnormalities; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Myelomonocytic, Chronic; Leukemia, Neutrophilic, Chronic; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelomonocytic, Juvenile; Lymphoma, B-Cell, Marginal Zone; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Burkitt Lymphoma; Hodgkin Disease; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Recurrence; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell | interventions — Filgrastim; Busulfan; Cyclophosphamide; Cyclosporine; Etoposide; Methotrexate; Radiotherapy

INTERVENTIONS:
Biological: filgrastim
Drug: busulfan
Drug: cyclophosphamide
Drug: cyclosporine
Drug: etoposide
Drug: methotrexate
Procedure: allogeneic bone marrow transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Giving chemotherapy drugs and total-body irradiation before a donor bone marrow transplant helps stop the growth of cancer and abnormal cells and helps stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Giving colony-stimulating factors, such as G-CSF, to the donor helps the stem cells move from the bone marrow to the blood so they can be collected and stored.

PURPOSE: This clinical trial is studying how well a G-CSF-treated donor bone marrow transplant works in treating patients with hematologic cancer or noncancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether granulocyte engraftment can be achieved by day 30 in patients with hematologic disorders undergoing HLA-matched, related-donor, allogeneic bone marrow transplantation using filgrastim (G-CSF)-primed bone marrow.
* Determine the incidence of grade II or greater acute graft-versus-host disease (GVHD) in patients treated with this regimen and post-transplantation immunosuppression with cyclosporine and methotrexate.

Secondary

* Determine whether platelet and red blood cell engraftment can be achieved in patients treated with this regimen.
* Determine the incidence of limited and extensive chronic GVHD in patients treated with this regimen.
* Determine the event-free survival of patients treated with this regimen.
* Determine the post-transplant immune reconstitution in patients treated with this regimen.

OUTLINE: This is a pilot study.

* Mobilization: Donors receive filgrastim (G-CSF) subcutaneously (SC) daily on days -3 to -1 followed by bone marrow collection.
* Conditioning regimen: Patients receive 1 of the following conditioning regimens according to their primary disease:

  * Total-body irradiation and high-dose chemotherapy comprising etoposide and cyclophosphamide
  * High-dose chemotherapy comprising busulfan and cyclophosphamide
* Bone marrow transplantation: Patients receive G-CSF-primed allogeneic bone marrow on day 0. Patients then receive G-CSF SC beginning on day 5.
* Graft-versus-host disease prophylaxis: Patients receive cyclosporine beginning on day -1 and methotrexate on days 1, 3, and 6.

PROJECTED ACCRUAL: A total of 15 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of hematologic malignancy or nonmalignancy
* Candidate for matched, related-donor, allogeneic bone marrow transplantation
* Availability of an HLA-matched (6/6) related donor

PATIENT CHARACTERISTICS:

Performance status

* ECOG 0-2 OR
* Karnofsky or Lansky 70-100%

Life expectancy

* At least 12 weeks

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* No significant functional deficit of any major organ

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior stem cell transplantation

Max Age: 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2004-05; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eneida Nemecek, MD, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States